CLINICAL TRIAL: NCT05150483
Title: EndotyPIng PreHospitAl de Novo Acute hYpoxemic Respiratory Failure
Acronym: EPIPHANY
Status: Recruiting | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Ilias Siempos, Assistant Professor in Critical Care and Pulmonary Medicine, Evangelismos Hospital
Other Study IDs: 80-1/15.10.2020
Record Dates: First submitted 2021-11-22; First posted 2021-12-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: critical illness; intensive care unit; endotypes; phenotypes; emergency department; trajectory; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Critical Illness; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with de novo acute hypoxemic respiratory failure: We will consider for inclusion patients presenting in the emergency department with de novo acute hypoxemic respiratory failure (AHRF). De novo AHRF is defined as the requirement of oxygen flow rate of 5 liters per minute or more to maintain SpO2 of 90% or more in a patient who does not receive long term oxygen therapy.

SUMMARY:
We attempt to perform dynamic endotyping of critically ill patients presenting in the emergency department with de novo acute hypoxemic respiratory failure (AHRF). We also attempt to identify what clinical, radiological, physiological and biological variables collected early in the course of AHRF correlate with subsequent mortality and/or persistent severe hypoxemia.

DETAILED DESCRIPTION:
Rationale:

Even before the pandemic of the new coronavirus disease (COVID-19), acute respiratory distress syndrome (ARDS), the most severe form of acute hypoxemic respiratory failure (AHRF), constituted a public health challenge. Despite the intense research on identifying targeted pharmacological therapies for ARDS, there is no available treatment for the syndrome.

The failure of clinical trials exploring pharmacological therapies for ARDS has been attributed to incomplete understanding of the pathogenesis and heterogeneity of the syndrome. As examples of the heterogeneity of ARDS, our recent work has identified differential outcomes of patients with ARDS depending on whether hypoxemia is rapidly improving or persistent severe or associated with non-identifiable risk factors or associated with neutropenia. It is advocated that the heterogeneity of ARDS can be tangled by a precision approach, which identifies endotypes of ARDS; i.e., subtypes characterized by a distinct biological profile that might share mortality risk, clinical course, or treatment responsiveness.

Notwithstanding their contributions, current research efforts on endotyping ARDS might be limited by the fact that they are based on the current conceptual framework of the syndrome, which has been widely questioned. Indeed, for reasons such as high interobserver variability of radiological criteria of ARDS and exclusion of patients requiring high-flow nasal oxygen, influential experts have even suggested to completely abandon the term.

Objective:

Accordingly, in the current study, we attempt to perform endotyping of critically ill patients presenting in the emergency department with de novo AHRF, which is a simpler and more reliable phenotype than ARDS. The approach for endotyping will be dynamic rather than static; i.e, two blood samples with a 24-hour interval will be used for endotyping to trace trajectories of biomarkers (over 1500 unique human proteins). In addition, we attempt to identify what clinical, radiological, physiological and biological variables collected early in the course of AHRF correlate with subsequent mortality and/or persistent severe hypoxemia.

Thus, the research protocol is organized as 3 aims.

Aim#1 will organize a registry and biobank of critically ill patients presenting in the emergency department with de novo AHRF.

Aim#2 will build a predictive model to identify what variables among those collected in Aim#1 are associated with subsequent mortality and/or persistent severe hypoxemia.

Aim#3 will use an agnostic discovery approach to explore novel proteomic biomarkers-based dynamic endotypes in critically ill patients presenting in the emergency department with de novo AHRF. Also, Aim#3 will create a multiprotein model of biomarkers associated with subsequent mortality and/or persistent severe hypoxemia and will determine whether inclusion of this multiprotein panel in the predictive score developed in Aim#2 improves risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >18 years) presenting in the emergency department
* De novo acute hypoxemic respiratory failure (requiring oxygen flow rate of 5 liters per minute or more to maintain SpO2 of 90% or more)

Exclusion Criteria:

* Age <18 years
* Not admitted to the hospital
* Postoperative acute respiratory failure (within one week from surgery)
* Chronic hypoxemic respiratory failure (requiring long term oxygen therapy at home)
* Hypercapnic respiratory failure
* Transferred from another hospital or facility
* Pregnant women
* Admitted to the hospital purely to facilitate comfort care
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting in the emergency department with de novo acute hypoxemic respiratory failure
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of dynamic endotypes of acute hypoxemic respiratory failure | Until death or hospital discharge, assessed up to 28 days following presentation to the emergency department
  Mutually exclusive subgroups of patients (clusters) characterized by a distinct biological profile that might share mortality risk, clinical course, and/or treatment responsiveness.

SECONDARY OUTCOMES:
All-cause mortality | Until death or hospital discharge, assessed up to 28 days following presentation to the emergency department
  To determine what variables among those collected, including protein biomarkers, are associated with subsequent all-cause mortality.
Persistent severe hypoxemia | Until 28 days following presentation to emergency department
  To determine what variables among those collected, including protein biomarkers, are associated with persistent severe hypoxemia. We will consider that persistent severe hypoxemia is present in endotracheally intubated individuals receiving positive pressure ventilation and having a PaO2:FiO2 ratio of equal to or less than 100 mmHg at 48 hours following intubation.
Intensive care unit-free days | Until 28 days following presentation to emergency department
  Intensive care unit-free days are calculated by the number of days in the first 28 days following presentation in the emergency department that a patient is alive and not in the intensive care unit.
Vasopressor-free days | Until 28 days following presentation to emergency department
  Vasopressor-free days are calculated by the number of days in the first 28 days following presentation in the emergency department that a patient is alive and not receiving vasopressors.
Ventilator-free days | Until 28 days following presentation to emergency department
  Ventilator-free days are calculated by the number of days in the first 28 days following presentation in the emergency department that a patient is alive and not on a ventilator.
Continuous renal replacement therapy-free days | Until 28 days following presentation to emergency department
  Continuous renal replacement therapy-free days are calculated by the number of days in the first 28 days following presentation in the emergency department that a patient is alive and not receiving continuous renal replacement therapy.
Bacteremia | Until 28 days following presentation to emergency department
  Bacteremia is determined by a positive blood culture.

CONTACTS AND LOCATIONS:
Overall Officials: Ilias I. Siempos, MD, DSc, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 3 months from publication
Access Criteria: For research use

REFERENCES:
- [Background] Meyer NJ, Gattinoni L, Calfee CS. Acute respiratory distress syndrome. Lancet. 2021 Aug 14;398(10300):622-637. doi: 10.1016/S0140-6736(21)00439-6. Epub 2021 Jul 1. PMID 34217425
- [Background] Beitler JR, Thompson BT, Baron RM, Bastarache JA, Denlinger LC, Esserman L, Gong MN, LaVange LM, Lewis RJ, Marshall JC, Martin TR, McAuley DF, Meyer NJ, Moss M, Reineck LA, Rubin E, Schmidt EP, Standiford TJ, Ware LB, Wong HR, Aggarwal NR, Calfee CS. Advancing precision medicine for acute respiratory distress syndrome. Lancet Respir Med. 2022 Jan;10(1):107-120. doi: 10.1016/S2213-2600(21)00157-0. Epub 2021 Jul 23. PMID 34310901
- [Background] Gattinoni L, Marini JJ. Isn't it time to abandon ARDS? The COVID-19 lesson. Crit Care. 2021 Sep 6;25(1):326. doi: 10.1186/s13054-021-03748-6. No abstract available. PMID 34488807
- [Background] Matthay MA, McAuley DF, Ware LB. Clinical trials in acute respiratory distress syndrome: challenges and opportunities. Lancet Respir Med. 2017 Jun;5(6):524-534. doi: 10.1016/S2213-2600(17)30188-1. Epub 2017 May 26. PMID 28664851
- [Background] Schenck EJ, Oromendia C, Torres LK, Berlin DA, Choi AMK, Siempos II. Rapidly Improving ARDS in Therapeutic Randomized Controlled Trials. Chest. 2019 Mar;155(3):474-482. doi: 10.1016/j.chest.2018.09.031. Epub 2018 Oct 22. PMID 30359616
- [Background] Sanchez E, Price DR, Chung KP, Oromendia C, Choi AMK, Schenck EJ, Siempos II. Persistent severe acute respiratory distress syndrome for the prognostic enrichment of trials. PLoS One. 2020 Jan 27;15(1):e0227346. doi: 10.1371/journal.pone.0227346. eCollection 2020. PMID 31986174
- [Background] Harrington JS, Schenck EJ, Oromendia C, Choi AMK, Siempos II. Acute respiratory distress syndrome without identifiable risk factors: A secondary analysis of the ARDS network trials. J Crit Care. 2018 Oct;47:49-54. doi: 10.1016/j.jcrc.2018.06.002. Epub 2018 Jun 2. PMID 29898428
- [Background] Price DR, Hoffman KL, Oromendia C, Torres LK, Schenck EJ, Choi ME, Choi AMK, Baron RM, Huh JW, Siempos II. Effect of Neutropenic Critical Illness on Development and Prognosis of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2021 Feb 15;203(4):504-508. doi: 10.1164/rccm.202003-0753LE. No abstract available. PMID 32986956